CLINICAL TRIAL: NCT05121376
Title: A Phase 1/2 Open-Label, Dose-Escalation Study to Determine the Safety Tolerability & Efficacy of BMN 331 an AAV Vector-Mediated Gene Transfer of Human SERPING1 Gene in Subjects With HAE Due to Human C1-INH Deficiency
Brief Title: A Gene Therapy Study of BMN 331 in Subjects With Hereditary Angioedema
Acronym: HAErmony-1
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 331-201
Record Dates: First submitted 2021-10-28; First posted 2021-11-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Hereditary Angioedema; HAE
Keywords: HAE; Hereditary Angioedema; Gene Therapy; 331-201; 331; Haermony
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMN 331 (Experimental): AAV Gene Therapy Infusion
  Interventions: Genetic: Dose 1 of BMN 331; Genetic: Dose 2 of BMN 331; Genetic: Dose 3 of BMN 331; Genetic: Dose 4 of BMN 331; Genetic: Dose 5 of BMN 331; Genetic: Dose 6 of BMN 331; Genetic: Dose 7 of BMN 331

INTERVENTIONS:
Genetic: Dose 1 of BMN 331 — BMN 331 AAV Gene Therapy
Genetic: Dose 2 of BMN 331 — BMN 331 AAV Gene Therapy
Genetic: Dose 3 of BMN 331 — BMN 331 AAV Gene Therapy
Genetic: Dose 4 of BMN 331 — BMN 331 AAV Gene Therapy
Genetic: Dose 5 of BMN 331 — BMN 331 AAV Gene Therapy
Genetic: Dose 6 of BMN 331 — BMN 331 AAV Gene Therapy
Genetic: Dose 7 of BMN 331 — BMN 331 AAV Gene Therapy

SUMMARY:
This is a Phase 1/2, single-arm, open-label, dose-escalation and dose-expansion study of BMN 331 for the treatment of hereditary angioedema (HAE) due to C1 Esterase Inhibitor (C1-INH) protein deficiency. The study drug BMN 331is identified as AAV5 hSERPING1, an adeno-associated virus (AAV5)-based gene therapy vector that expresses wild-type human C1 Esterase Inhibitor (hC1-INH), under the control of a liver-selective promoter, and is being developed for the treatment of HAE with C1-INH deficiency. The pharmaceutical form of BMN 331 is a solution for intravenous infusion.

DETAILED DESCRIPTION:
BMN 331 is an investigational, single administration gene therapy intended to modify the disease course of HAE. Preclinical studies have shown that BMN 331 can transduce hepatocytes resulting in restoration of the deficient circulating levels of hC1-INH that cause HAE.

Study 331-201 is a two-part (part A and part B), first-in-human, Phase 1/2 study designed to assess the safety and efficacy of BMN 331 in patients with HAE. Subjects will be followed for 5 years following BMN 331 infusion. Part A of the study is a dose escalation phase designed to assess the preliminary safety of a single IV administration of BMN 331 and to determine whether there is a dose-dependent increase in C1-INH protein expression following administration of BMN 331. Part B is a dose expansion phase designed to demonstrate that up to three safe doses of BMN 331 (as determined in Part A) sustains a clinically meaningful increase in C1-INH levels.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male adults ( ≥ 18 years old)
2. Part A only: Confirmed diagnosis of Type I HAE due to C1-INH deficiency confirmed by genotyping of the SERPING1 gene Part B only: Confirmed diagnosis of Type I or II HAE due to C1-INH deficiency confirmed by genotyping of the SERPING1 gene
3. Currently using an HAE medication regimen that consists of a routine long-term prophylactic treatment for at least 6 months prior to enrollment or an on-demand therapy regimen for a documented attack frequency of at least 4 attacks within the last 12 months prior to enrollment or at least 2 attacks within the last 6 months prior to enrollment
4. Trained in self-administering acute attack treatment and is able to adequately manage acute attacks in a home setting
5. Willingness to abstain from consumption of alcohol for at least 52 weeks post BMN 331 infusion and to use highly effective contraception

Exclusion Criteria:

1. Evidence of active or chronic infection, including severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), or any immunosuppressive disorder
2. Contraindication to using glucocorticosteroids GCS, including a diagnosis of glaucoma or untreated osteoporosis
3. Active malignancy (except non-melanoma skin cancer) autoimmune, metabolic (i.e., diabetes), hematologic, cardiac, or renal disease that is of clinical significance defined as requiring regular medical attention and treatment
4. Prior gene therapy treatment
5. Prior use of high-dose attenuated androgens in the last 1 year prior to the study
6. History or current clinically relevant liver disease (eg, nonalcoholic steatohepatitis [NASH], or chronic viral hepatitis B or C [HBV or HCV] or autoimmune hepatitis)
7. Have a history or are at risk for clinically significant thromboembolic events (TEE) , or known underlying risk factor for thrombosis including thrombotic microangiopathy (TMA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events following a single IV administration of BMN 331 | At 5 years
  Number of participants with treatment-emergent adverse events following a single IV administration of BMN 331

SECONDARY OUTCOMES:
Time-normalized number of investigator-confirmed HAE attacks | At 5 years
Time-normalized number of investigator-confirmed HAE attacks by severity (mild, moderate, severe) | At 5 years
Time-normalized use of HAE-specific medication | At 5 years
Plasma levels of functional C1-INH following BMN-331 infusion and change from baseline | At 5 years
Plasma levels of C1-INH antigen following BMN 331 infusion and change from baseline | At 5 years
Detection of total antibodies against AAV5 capsid following BMN 331 infusion | At 5 years
Detection of total antibodies against C1-INH following BMN 331 infusion | At 5 years
Detection of neutralizing antibodies against C1-INH following BMN 331 infusion | At 5 years

CONTACTS AND LOCATIONS:
Overall Officials: MD Medical Director, Study Director — BioMarin Pharmaceutical
Locations (16):
- United States (13):
  - AllerVie Clinical Research, Birmingham, Alabama
  - Medical Research of Arizona, Scottsdale, Arizona
  - University of California San Diego, San Diego, California
  - Asthma & Allergy Associates P.C., Colorado Springs, Colorado
  - Dr. Henry J. Kanarek Allergy, Asthma & Immunology, Overland Park, Kansas
  - Institute For Asthma & Allergy, Chevy Chase, Maryland
  - Mississippi Center for Advanced Medicine, Madison, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Duke Health, Durham, North Carolina
  - University of Cincinnati (UC) Physicians Company, LLC, Cincinnati, Ohio
  - Optimed Research, LTD, Columbus, Ohio
  - The Pennsylvania State University (Penn State) Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - AARA Research Center, Dallas, Texas
- Royal Prince Alfred Hospital,, Camperdown, Australia
- Spain (2):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid